CLINICAL TRIAL: NCT06914323
Title: The Effects of Acupressure on Pain, Swelling and Comfort in Patients With Femoral Fracture Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Yu-Tzu Chang, Nurse practitioner, Hungkuang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2025-03-11; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acupressure
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acupressure (Experimental)
  Interventions: Procedure: Acupressure

INTERVENTIONS:
Procedure: Acupressure — improvements in pain, limb swelling, and comfort

SUMMARY:
Pain is a subjective and unpleasant sensory and emotional experience associated with actual or potential tissue damage. Fractures result from a disruption in the continuity of bone, where bones are subjected to traction, twisting, or compression, causing damage to the surrounding muscular tissues. The treatment of displaced or complex fractures typically requires internal fixation surgery. 89% of fracture patients experience postoperative pain and swelling by the second day following open reduction and internal fixation surgery. These negative sensations can lead to increased pain, limb deformity, and neurovascular compression injuries. If postoperative pain is not adequately managed, it can affect wound healing, increase metabolism and oxygen consumption, and place additional strain on cardiopulmonary function. It is necessary to integrate alternative, non-pharmacological, non-invasive pain relief measures. Effectively and safely alleviating acute postoperative pain can enhance comfort, promote early mobilization, improve adherence to postoperative physical therapy, enhance quality of life and shorten hospital stays.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was hospitalized due to injuries from an accident, diagnosed with unilateral femoral fracture and underwent open reduction internal fixation surgery, hemiarthroplasty, and total hip arthroplasty.
2. Adults aged 18 years or older.
3. Conscious and able to communicate in Mandarin or Taiwanese (Min Nan).
4. Intact and without missing lower limbs.
5. Willing to sign the informed consent form after being briefed on the study objectives and procedures.

Exclusion Criteria:

1. Diagnosis of musculoskeletal tumors.
2. History of cerebrovascular accident or peripheral vascular neuropathy.
3. Major medical conditions such as cirrhosis, renal failure, heart failure, cancer, and severe brain diseases.
4. Edema caused by nutritional deficiency or mucinous causes.
5. Pregnant or lactating women.
6. Patients using patient-controlled analgesia post-surgery.
7. Severe psychiatric disorders or perceptual disorders.
8. Platelet count less than 20 x 10^3/uL before screening.
9. Albumin less than 3.5g/dL before screening.
10. Individuals closely related to the trial personnel, such as immediate family or dependents of the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Changes in pain | post op day 1 to post op day 2
  Pain is measured using the Visual Analog Scale (VAS). The left end is labeled as "no pain," which represents 0, and the right end as "the most severe pain imaginable," which represents 100.
Change in limb swelling | post op day 1 to post op day 2
  Foot circumference at the midpoint of the line connecting the fifth toe to the lateral malleola is measured in centimeters for swelling assessment. A measuring tape is used. During the measurement, the patient is positioned in a supine posture.
Changes in patient comfort | post op day 1 to post op day 2
  Shortened General Comfort Questionnaire (SGCQ) for measuring comfort. The questionnaire consists of 28 items, assessed on a 6-point Likert scale ranging from "strongly disagree" to "strongly agree." A score of 1 represents "strongly disagree," while a score of 6 represents "strongly agree." The total score ranges from 28 to 148, with higher scores indicating greater levels of comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Hungkuang University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No